CLINICAL TRIAL: NCT05443867
Title: Monkeypox ASymptomatic Shedding: Evaluation by Self-Sampling MPX-ASSESS
Acronym: MPX-Assess
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: MPX-Assess
Record Dates: First submitted 2022-06-21; First posted 2022-07-05 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Monkey Pox
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood
  * Oropharyngeal swab
  * Anal swab (self-sampling)
  * Genital swab (self-sampling)
  * Saliva (self-sampling)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MPX-Assess: Contacts of MPX index cases

SUMMARY:
Monkeypox (MPX) is a viral zoonosis, caused by the Monkeypox virus (MPXV), a DNA virus that belongs to the Orthopoxvirus genus and is closely related to the variola virus, the causative agent of smallpox. Until recently the spread of MPX was mainly confined to the Central African rainforest and to parts of West Africa. However, in May 2022, several cases of MPX were detected throughout Europe and Northern America, albeit with a different presentation than previously seen. Many questions remain on this new presentation of the disease: what the exact mode of transmission is, how contagious the virus really is and whether asymptomatic carriers exist. With this study the researchers aim to perform a close follow-up study of close contacts of MPX confirmed cases. Participants are recruited among high and very high risk contacts of confirmed monkeypox patients that presented to the ITM for diagnosis (index). Contacts that are asymptomatic (for symptoms compatible with MPXV infection according to national case definitions) at the time of recruitment will be enrolled. Contacts of the index case that are symptomatic at recruitment or become symptomatic during follow-up will be invited for sample collection at different timepoints until 21 days after contact as suspect cases.

ELIGIBILITY:
Inclusion Criteria:

1. Be a high risk or very high-risk contact of a laboratory confirmed monkeypox case, with:

   * Very high-risk contact:

     * Sexual partner(s)
     * Prolonged skin-to-skin contact while the patient had skin lesions
   * High risk contact

     * living in the same household or similar environment (e.g. camping, spending the night, etc.);
     * shared clothing, bedding, utensils, etc., while the patient had skin lesions
     * healthcare workers with unprotected contact (inadequate or no PPE)
2. Last exposure to the monkeypox index case of less than 21 days ago
3. Adult participants (≥ 18 years old) of any gender
4. Written informed consent is obtained from the participant

Exclusion Criteria:

1. Presenting with symptoms compatible with MPX:

   * an unexplained rash on any part of the body AND
   * one or more of the following symptoms: fever, headache, back pain, fatigue, lymphadenopathy (localised or generalised)
2. Inability or unwillingness to comply with the proposed follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are recruited among high and very high risk contacts of confirmed monkeypox patients that presented to the ITM for diagnosis (index). Contacts that are asymptomatic (for symptoms compatible with MPXV infection according to national case definitions) at the time of recruitment will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Secondary attack rate of MPXV infection in contacts, defined by PCR positivity on any sample | Until 21 days after contact with index case
  Secondary attack rate of MPXV infection in contacts, defined by PCR positivity on any sample

SECONDARY OUTCOMES:
Rate of seroconversion in contacts, defined as a positive IgG (immunoglobulineG) for monkeypox | Until 21 days after contact with index case
  To evaluate the rate of seroconversion in contacts (positive IgG for MPX) within 21 days after contact with index case
Proportion of seroconversion in PCR positive contacts vs PCR negative contacts, defined as negative MPXV PCR in all samples until the end of the follow-up period | Until 21 days after contact with index case
  Proportion of seroconversion in PCR positive contacts vs PCR negative contacts, defined as negative MPXV PCR in all samples until the end of the follow-up period
Time to seroconversion overall, in symptomatic and asymptomatic contacts, and in PCR positive and negative cases | Until 21 days after contact with index case
  Time to seroconversion overall, in symptomatic and asymptomatic contacts, and in PCR positive and negative cases
Proportion of PCR positive participants with asymptomatic infection at time of first positive PCR | Until 21 days after contact with index case
  Proportion of PCR positive participants with asymptomatic infection at time of first positive PCR
Proportion of PCR positive participants developing symptoms within the follow-up period | Until 21 days after contact with index case
  Proportion of PCR positive participants developing symptoms within the follow-up period
Proportion of asymptomatic infections on number of contacts in follow-up. Asymptomatic infections are defined as contacts with positive MPXV PCR on any clinical sample, without development of any symptoms. | within 3 weeks after exposure or within 1 week after PCR positivity, whichever follow-up is longer
  Proportion of asymptomatic infections on number of contacts in follow-up. Asymptomatic infections are defined as contacts with positive MPXV PCR on any clinical sample, without development of any symptoms within 3 weeks after exposure or within 1 week after PCR positivity, whichever follow-up is longer
Time from MPXV PCR positivity in any sample to appearance of any symptom overall and per mode of transmission (close personal contact; anal, vaginal or oral receptive sexual contact; and insertive sexual contact) | at the end of the 3-week follow-up period
  Time from MPXV PCR positivity in any sample to appearance of any symptom overall and per mode of transmission (close personal contact; anal, vaginal or oral receptive sexual contact; and insertive sexual contact)
Time from MPXV PCR positivity in any sample to appearance of skin lesions | at the end of the 3-week follow-up period
  Time from MPXV PCR positivity in any sample to appearance of skin lesions
Time from confirmed exposure to first PCR positivity | at the end of the 3-week follow-up period
  Time from confirmed exposure to first PCR positivity
Time from confirmed exposure to appearance of any symptom | at the end of the 3-week follow-up period
  Time from confirmed exposure to appearance of any symptom
Time from confirmed exposure to appearance of skin lesions | at the end of the 3-week follow-up period
  Time from confirmed exposure to appearance of skin lesions
Description of the type of symptoms observed in monkeypox contacts | within 3 weeks after last exposure
  Description of the type of symptoms observed in monkeypox contacts within 3 weeks after last exposure
Frequency of symptoms observed in monkeypox contacts | within 3 weeks after last exposure
  Frequency of symptoms observed in monkeypox contacts within 3 weeks after last exposure
Timing of symptoms observed in monkeypox contacts | within 3 weeks after last exposure
  Timing of symptoms observed in monkeypox contacts within 3 weeks after last exposure
Distribution of skin lesions for sexual contacts versus close personal contacts. (per body surface and per category: local vs generalized skin lesions) | at the end of the 3-week follow-up period
  Distribution of skin lesions for sexual contacts versus close personal contacts. (per body surface and per category: local vs generalized skin lesions)
Proportion of contacts presenting with systemic symptoms after sexual exposure versus those with close personal contacts exposure | at the end of the 3-week follow-up period
  Proportion of contacts presenting with systemic symptoms after sexual exposure versus those with close personal contacts exposure
Number of contacts with the defined risk and protective factors | At baseline
  Number of contacts with the defined risk and protective factors
Proportion of presence of defined factors in PCR positive contacts. | Until the end of the 3-week follow-up period
  Proportion of presence of defined factors in PCR positive contacts.
Proportion of presence of defined factors in symptomatic PCR positive contacts | Until the end of the 3-week follow-up period
  Proportion of presence of defined factors in symptomatic PCR positive contacts

OTHER OUTCOMES:
Presence of culturable virus in PCR positive samples from pre- or asymptomatic period | Until the end of the 3-week follow-up period
  Presence of culturable virus in PCR positive samples from pre- or asymptomatic period

CONTACTS AND LOCATIONS:
Overall Officials: Laurens Liesenborghs, MD, Principal Investigator — Instituut van Tropische Geneeskunde Antwerpen
Locations (1):
- Institute of Tropical Medicine Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Brosius I, Van Dijck C, Coppens J, Vandenhove L, Bangwen E, Vanroye F, Verschueren J; ITM MPOX Study Group; Zange S, Bugert J, Michiels J, Bottieau E, Soentjens P, van Griensven J, Kenyon C, Arien KK, Van Esbroeck M, Vercauteren K, Liesenborghs L. Presymptomatic viral shedding in high-risk mpox contacts: A prospective cohort study. J Med Virol. 2023 May;95(5):e28769. doi: 10.1002/jmv.28769. PMID 37212312